CLINICAL TRIAL: NCT02426710
Title: The Usefulness of Intracardiac Echocardiography in Atrial Flutter Ablation - a Randomized Study
Brief Title: Intracardiac Echocardiography in Atrial Flutter Ablation
Acronym: FLS-ICE-R
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Pavel Osmancik, Cardiocenter, III rd internal-cardiology clinic, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLS-ICE randomized
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: ATRIAL FLUTTER
Keywords: ablation, atrial flutter, intracardiac echocardiography
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Intervention Model Description: RAndomization to ICE or no ICE
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flutter ablation with intracardiac echocardiography (Experimental): Atrial flutter ablation will be done using intracardiac echocardiography.
  Interventions: Device: Intracardiac echocardiography
- Flutter ablation without intracardiac echocardiography (Active Comparator): Atrial flutter ablation will be done without intracardiac echocardiography.
  Interventions: Device: Intracardiac echocardiography

INTERVENTIONS:
Device: Intracardiac echocardiography — Flutter ablation will be done using intracardiac echocardiography.

SUMMARY:
Background: Radiofrequency ablation of typical atrial flutter present the most effective treament option in treatment of atrial flutter. Despite its high efficacy, due tovariant anatomy of cavotricuspid isthmus (CTI), i.e. location of right coronary artery, pouches, the achievment of complete bidirectional block across the CTI is sometimes chalenging. Intracardiac echocardiography (ICE) is a very usefull tool for on-line vizualization of the anatomy of the atria and also for the location of catheter position on CTI during ablation. If the routine use of ICE is associated with easier atrial fluter ablation is not clear.

Methods: One hundred consecutive patients indicated for typical atrial flutter ablation will be enrolled into the study. The patients will be randomized into group (A) ablation with use of ICE and (B) ablation without ICE. The ablation will be done in both groups by two diagnostic catheters (10-pole positioned in coronary sinus and 20-pole halo catheter positioned in the right atrium) and radiofrequency ablation catheter. The end-point of the ablation is the achievment of the bicidrectional block across the CTI. The end-points of the study are 1) the total length of the procedure, 2) the fluoroscopy time and 3) the ablation time. The safety end-point is clinically significant bleeding from the groin due to additional puncture for ICE catheter.

Discussion: We hypothesize the use of ICE wil shorten the radiofrequency energy delivery, fluoroscopy time and the length of the procedure without increasing the bleeding.

DETAILED DESCRIPTION:
Introduction Radiofrequency ablation (RFA) of typical atrial flutteru is the most successful method for treatment of atrial flutter. The acute (peri-procedural) efficacy is more than 95%. (1) Typical atrial flutter circuit uses the area between inferior caval vein and tricuspid anulus, so a RFA of typical flutter is performed by providing a linear lesion from inferior caval vein to tricuspid valve (this area is called as cavo-tricuspid isthmus). The recurrence of atrial flutter after ablation, which are caused by non-transmural RF lesion, are in less than 10% of cases. (2) During atrial flutter ablation, typically three electrophysiological catheters are used. Two catheters are diagnostic (one 10-pole inserted into coronary sinus and the other 20-pole inserted in the right atrium with the distal tip laterally from the cavo-ticuspid isthmus). The third is ablation catheter, inserted in the CT isthmus. The location of all three catheters is monitored by fluoroscopy and by the EP signals on catheters. Also the ablation catheter during the ablation is monitored by fluoroscopy and by the signals on the catheter.

Despite its high efficacy, the RFA of atrial flutter can be sometimes very difficult. The most difficulties are done by anatomical differences in patients. (3, 4) In the area of CTI, the rudimentary Eustachian valve can be present, which can hide the effective ablation of the CI tissue. Moreover, deep pouches can be present in the TI area, which, if unrecognized, can present the area of insufficient ablation. Both of them, Eustachian valve or pouches, are not visible by fluoroscopy. In rare cases, a complete block in the CTI are is not achieved, typically due to some anatomical difficulties. Furthermore, this anatomical obstacles can lead to prolonged fluoroscopy time (to find the location of conduction in CTI rea), more RF energy delivery and prolonged procedure time. Longer ablation time increases the risk of ablation (such as right atrial perforation). Next possible anatomical obstacle is the right coronary artery which can effective prevent sufficient ablation due to its cooling effect. (5) Intracardiac echocardiography (ICE) is done by using intracardiac echo probe. The probe is inserted in the right atrium, which allows the visualizing of the CTI area. (6, 7) ICE is used for AF ablation in some centers, but its effect has never been validated in the randomized study. The aim of our study is to assess whether routine use of ICE can lead to decrease fluoroscopy time, decrease need for RFA delivery (i.e. number of ablations) and a decrease procedure time. On the other hand, the safety endpoint will be to assess whether a routine use of ICE is not associated with higher rate of complications. We hypothesize, the use of ICE will shorten fluoroscopy, ablation and procedural time without increased number of complication

Patients and methods:

Consecutive patients indicated due to standard criteria (i.e. according to the guidelines of the European Society of Cardiology) for atrial flutter ablation will be enrolled. Exclusion criterion will be the absence of written informed content and a history of recent femoral vein thrombosis (< 6 months).

Randomization: 1 to 1 for ICE vs. non ICE RF ablation will be done routinely, as it is done in the center. In the Ice group, ICE probe will be inserted through the left femoral vein in the right atrium TH ICE will be used for the visualization of the anatomy of CTI area and the visualization of the catheter during RF delivery. In case of the non-ICE group, RFA will be done without ICE catheter, as it is done routinely now. In both groups, the diagnostic catheters (10-pole CS and 20-po in the RA) and ablation catheter will be the same. In the non-ICE group, the location of the catheters will be assessed by fluoroscopy and by signals on catheters. At the end of ablation, total fluoroscopy time, the number and length of ablation and the duration of procedure will be calculated. On the day and two weeks after the procedure, the bleeding complication will be assessed.

End-points: the major end-points will be: 1) total procedure duration (min) 2) fluoroscopy time 3) the number of ablations 4) the total duration of RF energy delivery. Major safety end-point will be complication from left femoral ICE access.

ELIGIBILITY:
Inclusion Criteria:

* indication for atrial flutter ablation

Exclusion Criteria:

* history of recent femoral vein thrombosis (within last 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-06; Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Procedure duration | intraoperative
  The total lenght of the procedure in minuts will be measured.
Fluoroscopy time during ablation | intraoperative
  The total fluoroscopy time will be measured.
Total ablation time | intraoperative
  The time of radiofrequenc energy delivery during ablation will me measured.
Bleeding | 24 hours
  The bleeding complication required intervention or prolonged hospitalization will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiocenter, 3rd Medical School, Charles University and University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
Study was published

REFERENCES:
- [Background] Scaglione M, Caponi D, Di Donna P, Riccardi R, Bocchiardo M, Azzaro G, Leuzzi S, Gaita F. Typical atrial flutter ablation outcome: correlation with isthmus anatomy using intracardiac echo 3D reconstruction. Europace. 2004 Sep;6(5):407-17. doi: 10.1016/j.eupc.2004.05.008. PMID 15294265
- [Result] Lee G, Sanders P, Kalman JM. Catheter ablation of atrial arrhythmias: state of the art. Lancet. 2012 Oct 27;380(9852):1509-19. doi: 10.1016/S0140-6736(12)61463-9. PMID 23101718
- [Result] Schumacher B, Pfeiffer D, Tebbenjohanns J, Lewalter T, Jung W, Luderitz B. Acute and long-term effects of consecutive radiofrequency applications on conduction properties of the subeustachian isthmus in type I atrial flutter. J Cardiovasc Electrophysiol. 1998 Feb;9(2):152-63. doi: 10.1111/j.1540-8167.1998.tb00896.x. PMID 9511889
- [Result] Gami AS, Edwards WD, Lachman N, Friedman PA, Talreja D, Munger TM, Hammill SC, Packer DL, Asirvatham SJ. Electrophysiological anatomy of typical atrial flutter: the posterior boundary and causes for difficulty with ablation. J Cardiovasc Electrophysiol. 2010 Feb;21(2):144-9. doi: 10.1111/j.1540-8167.2009.01607.x. Epub 2009 Oct 5. PMID 19804553
- [Result] Lai LP, Lin JL, Lin JM, Du CC, Tseng YZ, Huang SK. Use of double-potential barrier to identify functional isthmus at the cavotricuspid isthmus for facilitating catheter ablation of isthmus-dependent atrial flutter. J Cardiovasc Electrophysiol. 2004 Apr;15(4):396-401. doi: 10.1046/j.1540-8167.2004.03424.x. PMID 15089986
- [Result] Al Aloul B, Sigurdsson G, Can I, Li JM, Dykoski R, Tholakanahalli VN. Proximity of right coronary artery to cavotricuspid isthmus as determined by computed tomography. Pacing Clin Electrophysiol. 2010 Nov;33(11):1319-23. doi: 10.1111/j.1540-8159.2010.02844.x. PMID 20663073
- [Result] Morton JB, Sanders P, Davidson NC, Sparks PB, Vohra JK, Kalman JM. Phased-array intracardiac echocardiography for defining cavotricuspid isthmus anatomy during radiofrequency ablation of typical atrial flutter. J Cardiovasc Electrophysiol. 2003 Jun;14(6):591-7. doi: 10.1046/j.1540-8167.2003.02152.x. PMID 12875419